CLINICAL TRIAL: NCT00976274
Title: Effects of Korean Red Ginseng on Cardiovascular Risks in Subjects With Metabolic Syndrome
Brief Title: Korean Red Ginseng and Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Korean Society of Ginseng (Other)
Responsible Party: Principal Investigator, Jae-Yong Shim, Professor, The Korean Society of Ginseng
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3-2009-0015
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Results first posted 2012-02-24 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-02

CONDITIONS: Metabolic Syndrome
Keywords: Korean red ginseng; metabolic syndrome; blood pressure; arterial stiffness; inflammation; oxidative stress
MeSH Terms: conditions — Metabolic Syndrome; Inflammation | interventions — Asian ginseng; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- starch capsule (Placebo Comparator)
  Interventions: Dietary Supplement: starch
- Korea red ginseng (Experimental)
  Interventions: Dietary Supplement: Korean red ginseng

INTERVENTIONS:
Dietary Supplement: Korean red ginseng — 5 capsules (300 mg/capsule) three times everyday for 12 weeks
  Other Names: Korean Red Ginseng Powder Capsule, KGC1039012
  Arms: Korea red ginseng
Dietary Supplement: starch — 5 capsules three times everyday for 12 weeks
  Other Names: KGC1039015
  Arms: starch capsule

SUMMARY:
Five factor consisting of Metabolic syndrome is closely linked by insulin resistance. Until now, several studies have been performed about effects of Korea red ginseng on hypertension, diabetes, and hyperlipidemia, but not metabolic syndrome.

The investigators hypothesize that Korean red ginseng could improve each constituents of metabolic syndrome, arterial stiffness, and inflammatory markers.

The aim of this study is to determine effects of Korean red ginseng on cardiovascular risks in subjects with metabolic syndrome.

DETAILED DESCRIPTION:
The details of study objective are followed by these:

* comparison of blood pressure before and after Korean red ginseng administration
* comparison of metabolic indicator before and after Korean red ginseng administration
* comparison of oxidative stress and inflammatory markers before and after Korean red ginseng administration
* comparison of arterial stiffness before and after Korean red ginseng administration

ELIGIBILITY:
Inclusion Criteria:(three or more of following five factors)

* waist circumference(male: more than 90cm, female: more than 80cm)
* blood pressure(systolic: more than 130mmHg, diastolic: more than 85mmHg)
* fasting plasma glucose: more than 100mg/dL
* fasting triglycerides: more than 150mg/dL
* High-density lipoprotein(HDL)-cholesterol(male: less than 40mg/dL, female: less than 50mg/dL)

Exclusion Criteria: (any one of following factors)

* uncontrolled blood pressure(systolic: more than 160mmHg, diastolic: more than 100mmHg) or subjects taking blood pressure lowering drug
* Type 2 diabetes patients or fasting plasma glucose more than 126mg/dL
* triglyceride more than 400mg/dL, total cholesterol more than 250mg/dL
* subjects taking antilipidemic drug
* past history of coronary heart disease or cerebrovascular disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Yong Shim, Ph.D., Principal Investigator — Yonsei University College of Medicine Gangnam severance Hospital
Locations (1):
- Yonsei Univeristy College of Medicine, Gangnam Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Park BJ, Lee YJ, Lee HR, Jung DH, Na HY, Kim HB, Shim JY. Effects of Korean Red Ginseng on Cardiovascular Risks in Subjects with Metabolic Syndrome: a Double-blind Randomized Controlled Study. Korean J Fam Med. 2012 Jul;33(4):190-6. doi: 10.4082/kjfm.2012.33.4.190. Epub 2012 Jul 25. PMID 22916320

RESULTS

PARTICIPANT FLOW:
Groups:
- Starch Capsule: 5 capsules three times everyday for 12 weeks
- Korea Red Ginseng: 5 capsules (300mg/capsule) three times everyday for 12 weeks
Period: Overall Study
Arm/Group | Starch Capsule | Korea Red Ginseng
Started | 31 | 29
Completed | 24 | 21
Not Completed | 7 | 8
Not completed — Lost to Follow-up | 5 | 5
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Physician Decision | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Starch Capsule | Korea Red Ginseng | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 28 | 57
  >=65 years | 2 | 1 | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 46.2 (11.0) | 43.1 (10.6) | 44.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 19 | 20 | 39
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 31 | 29 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in the Pre- and Post-treatment Systolic Blood Pressure
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Starch Capsule | Korea Red Ginseng
Number analyzed (Participants) | 24 | 21
mm Hg
  Week 0 | 129.5 (10.7) | 134.5 (12.5)
  Week 12 | 122.6 (13.2) | 127.5 (13.6)

2. Secondary Outcome: Change in the Pre- and Post-treatment Oxidized Low-densty Lipoprotein(LDL)
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: uIU/mL
Arm/Group | Starch Capsule | Korea Red Ginseng
Number analyzed (Participants) | 24 | 21
uIU/mL
  0 week | 83.3 (35.9) | 78.8 (37.2)
  12 week | 83.4 (36.7) | 76.3 (29.0)

ADVERSE EVENTS:
Arm/Group | Starch Capsule | Korea Red Ginseng
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29
Other Adverse Events (participants affected / at risk) | 0/31 | 0/29

LIMITATIONS AND CAVEATS:
First, we could not fully control participants' lifestyle such as exercise and diet.Second, the relationship between Korean red ginseng dosage and its effect on cardiovascular disease risks was not evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No